CLINICAL TRIAL: NCT02133261
Title: BDx 7 Day ECG Patch: Electrode Adhesion Clinical Study
Status: Completed | Type: Observational
Sponsor: Bardy Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 7 day study
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Cardiac Patients; ECG Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to learn if a new 7 day patch ECG recording monitor can serve the same purpose as standard monitoring systems. The new 7day patch is significantly smaller and lighter than previous ECG recorders.

DETAILED DESCRIPTION:
The primary purpose of this research is to evaluate ECG signal quality of the BDx 7 day ECG Patch heart monitor after 7 full days of wear, establishing that the device is safe and effective to wear for up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* cardiac patient volunteers (5 male and 5 female)

Exclusion Criteria:

* skin rash or infection over the sternum
* Sternal incision within 3 months from the date of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac patients followed at the study site's location
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
adhesive performance/durability | 7 days
  The study will evaluate adhesive performance/durability by evaluating the Signal Quality of ECG data on the subjects (5 men and 5 women) in accordance with the requirements of FDA's ECG Electrode Guidance (section 5.A.3)1 and the ANSI/AAMI EC-12 Disposable ECG electrode technical standard (sections 4.4 and 5.4)2.

SECONDARY OUTCOMES:
human factors | 7 days
  Skin comfort or discomfort Device comfort Device stability and contact

CONTACTS AND LOCATIONS:
Overall Officials: Gene Trobaugh, MD, Principal Investigator — EvergreenHealth
Locations (1):
- EvergreenHealth, Enumclaw, Washington, United States